CLINICAL TRIAL: NCT00766948
Title: The Parkinson's Disease NeuroGenebank at Scripps Clinic Registry
Status: Active, not recruiting | Type: Observational
Sponsor: Scripps Translational Science Institute (Other)
Collaborators: Scripps Health (Other); The Scripps Research Institute (Other)
Responsible Party: Principal Investigator, Eric Topol, MD, Director, Scripps Translational Science Institute
Other Study IDs: HSC# 08-5022
Record Dates: First submitted 2008-10-02; First posted 2008-10-06 (Estimated); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood or Saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No Treatment
  Interventions: Other: There is no intervention, this is a biorepository.

INTERVENTIONS:
Other: There is no intervention, this is a biorepository. — There are no interventions in this study.

SUMMARY:
By creating a neurogenebank from Parkinson's disease patients' blood donations we will ultimately be able to define genes for Parkinson's disease and other neurological conditions.

ELIGIBILITY:
Inclusion Criteria:

* Is age 30 years or older at the time of onset of Parkinson's
* Has been diagnosed with idiopathic Parkinson's Disease by a Scripps Neurologist
* Is reliable, cooperative and willing to comply with all protocol-specified procedures and/or sub-study if consented or have legal representative/guardian willing to do so
* Able to understand and grant informed consent or have a legal representative/ guardian who is able to do so

Exclusion Criteria:

* Patient has been previously enrolled in The Parkinson's Disease NeuroGenebank at Scripps Clinic Registry
* If a blood draw would be contraindicated for any reason
* Has a significant chronic medical condition (i.e. CVA, hepatic encephalopathy) which, in the investigator's option, may interfere with the patient's optimal participation in the study
* Treatment with any investigational agents or devices within 30 days preceding enrollment in the study
* Has undergone ECT within 90 days preceding enrollment in the study

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 30 years of age or older with the diagnosis idiopathic Parkinson's disease
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-08; Primary Completion 2030-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Neurogenetic databank | Study completion
  initiate a Parkinson's disease neurogenetic databank by obtaining blood samples in order to define genes for Parkinson's disease and other neurological conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Cinnamon Bloss, PhD, Principal Investigator — Scripps Translational Science Institute and Genomic Medicine
Locations (3):
- United States (3):
  - Scripps Clinic, Torrey Pines, La Jolla, California
  - Scripps Translational Science Institute, La Jolla, California
  - The Scripps Research Institute, La Jolla, California